CLINICAL TRIAL: NCT04132726
Title: Effect of Massage Treatment in Patients With Temporomandibular Disorder
Brief Title: Effect of Massage Treatment in Temporomandibular Joint
Acronym: TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Merve Benli, Asst.Prof.Dr., Istanbul University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 192021
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Massage Therapy; Temporomandibular Disorder
Keywords: Massage
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test (Experimental): Experimental group which employed with massage treatment
  Interventions: Other: Massage therapy
- Placebo (Placebo Comparator): Placebo group which employed with non-effective treatment
  Interventions: Other: non-effective treatment
- Control (No Intervention): no treatment

INTERVENTIONS:
Other: Massage therapy — Massage therapy performed by a physiotherapist
  Arms: Test
Other: non-effective treatment — non-effective treatment
  Arms: Placebo

SUMMARY:
Temporomandibular disorders (TMD) have multiple and broad clinical effects on orofacial structures and are often diagnosed in patients with a prevalence of between 5% and 12%. Among treatment options, massage therapy is one of the common therapeutic procedures and allows interesting clinical outcomes by reducing TMD symptoms successfully. However, there has been no attempt to validate this knowledge. Thus, the aim of this study is to evaluate the effect of massage and its properties in patients with TMD.

ELIGIBILITY:
Inclusion Criteria:

1. Temporomandibular disorder-positive RDC/TMD examination for groups RDC/TMD Ia and RDC/TMD Ib,
2. Patient agreement to participate in the experimental study.

Exclusion Criteria:

1. RDC/TMD II and RDC/TMDIII,
2. Drug and/or removable partial or total prosthesis wearers,
3. Being submitted to any type of physiotherapeutic treatment,
4. Incomplete dentition,
5. History of systemic diseases as diabetes or arthritis,
6. The occurrence of facial trauma,
7. Refusal to assume responsibility with this research.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Pain- Visual Analog Scale | 12 weeks-14 weeks
  Self-reported pain values. High scores for pain mean worse outcome for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Benli, Dr., Principal Investigator — Istanbul University
Locations (1):
- Istanbul university,Faculty of Dentistry, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Capellini VK, de Souza GS, de Faria CR. Massage therapy in the management of myogenic TMD: a pilot study. J Appl Oral Sci. 2006 Jan;14(1):21-6. doi: 10.1590/s1678-77572006000100005. PMID 19089025